CLINICAL TRIAL: NCT03279146
Title: Open-Label, Part-Randomized Study Designed to Evaluate the PK Profile of Tenofovir Exalidex (TXL) Following Single Dose of Oral Formulations in Comparison to a Reference IR TXL Tablet in Healthy Subjects
Brief Title: A Single Dose Study Evaluating PK of TXL Oral Formulations in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ContraVir Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: ContraVir (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CTRV-TXL-103
Record Dates: First submitted 2017-08-18; First posted 2017-09-12 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Drug: Tenofovir Exalidex (TXL) oral formulations Other names: Lipid conjugateTFV
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Regimen A (Active Comparator): Immediate release tablet Tenofovir exalidex (TXL)
  Interventions: Drug: Tenofovir exalidex (TXL)
- Regimen B (Experimental): New Formulation 1 Tenofovir exalidex (TXL)
  Interventions: Drug: Tenofovir exalidex (TXL)
- Regimen C (Experimental): New formulation 2 Tenofovir exalidex (TXL)
  Interventions: Drug: Tenofovir exalidex (TXL)

INTERVENTIONS:
Drug: Tenofovir exalidex (TXL) — Oral formulations
  Other Names: Lipid conjugate YTFV

SUMMARY:
This is a Phase 1 study to evaluate the PK profile of TXL oral formulations in healthy subjects

DETAILED DESCRIPTION:
This is a Phase 1 study to evaluate the PK profile of different oral formulations of TXL following single dose administration in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-55 Capable of giving written informed consent Capable of completing study requirements

Exclusion Criteria:

* History or medical condition which could impact patient safety History of drug or alcohol abuse within past 2 years Positive result for HIV, HBV, or HCV Participation in another clinical trial within the past 90 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-06-09 (Actual); Study Completion 2018-06-16 (Actual)

PRIMARY OUTCOMES:
Evaluation of pharmacokinetics of single dose oral formulations of TXL in fasted state | up to four days post dose
  Measuring Cmax, the peak plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: John Sullivan-Bolyai, MD, MPH, Study Chair — ContraVir Pharmaceuticals
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided